CLINICAL TRIAL: NCT06231017
Title: A Single-arm, Open-label, Phase Ⅱ Clinical Trial of Adebrelimab Plus Cetuximab and Chemotherapy for Patients With RAS/BRAF Wild-Type Unresectable Liver Metastases Colorectal Cancer
Brief Title: Adebrelimab Plus Cetuximab and Chemotherapy for Patients With RAS/BRAF Wild-Type Unresectable Liver Metastases Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hong Zong, A Single-arm, Open-label, Phase Ⅱ Clinical Trial of Adebrelimab Plus Cetuximab and Chemotherapy for Patients With RAS/BRAF Wild-Type Unresectable Liver Metastases Colorectal Cancer, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2023-K019-003
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab + Cetuximab+ Chemotherapy (Experimental): Adebrelimab + Cetuximab+ Chemotherapy
  Interventions: Drug: Adebrelimab + Cetuximab+ Chemotherapy

INTERVENTIONS:
Drug: Adebrelimab + Cetuximab+ Chemotherapy — Adebrelimab:1200 mg, D1, Q2W+Cetuximab:500 mg, D1, Q2W+FOLFOX6(Q2W) or FOLFIRI(Q2W) until PD or resectability or to max 12 cycles

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of adebrelimab plus cetuximab and chemotherapy for patients with RAS/BRAF wild-type unresectable liver metastases colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is the third largest malignant tumor in the world and a significant cause of cancer-related deaths. The probability of simultaneous liver metastasis in colorectal cancer is about 25%, and the proportion of liver metastasis occurring in the entire disease process is as high as 40% -50%. It is of great clinical significance to transform the initial unresectable liver metastases of colorectal cancer into resectable ones to improve the overall survival rate and prognosis of colorectal cancer patients. We designed a single-arm, open phase II clinical trial of adebrelimab plus cetuximab and chemotherapy for patients with RAS/BRAF wild-type unresectable liver metastases colorectal cancer. The purpose of this study is to observe and evaluate the efficacy and safety of adebrelimab plus cetuximab and chemotherapy for patients with RAS/BRAF wild-type unresectable liver metastases colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have fully understood and voluntarily signed informed consent forms for this study, have good compliance, and cooperate with follow-up; 2. Age ≥ 18 years and ≤ 75 years old; 3. ECOG 0-1; 4. Expected survival time ≥ 12 weeks; 5. Patients confirmed by histology or pathology to have colon or rectal glands; 6. Primary or metastatic tumors of the colon are identified as RAS/BRAF wild-type; 7. PET/CT scan, CT scan, MRI or intraoperative exploration diagnosis (if applicable during resection of primary colorectal tumor), record evidence of limited liver metastasis in the patient (histological confirmation of liver metastasis is not required); 8. Primary colorectal cancer can be or has been radically resected, initial inability to R0 resection of liver metastases, or residual liver volume ≤ 30-40% after resection; 9. The patient has at least one measurable liver metastasis lesion (according to RECIST 1.1 standard); 10. There was no previous liver metastasis chemotherapy; 11. The main organ function is normal, which meets the following criteria:

1. Blood routine examination criteria should be met (no blood transfusion and blood products within 14 days, no correction with G-CSF and other hematopoietic stimulating factors):

   A. Hemoglobin (Hb) ≥ 90 g/L; B. Neutrophil count (ANC) ≥ 1.5 × 109/L; C. Platelet count (PLT) ≥ 100 × 109/L;
2. Biochemical examination must meet the following standards:

   A. Total bilirubin (TBIL)<1.5 upper limit of normal value (ULN); B. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are less than 2.5 ULN, while for patients with liver metastasis, they are less than 5 ULN; C. Serum creatinine (Cr) ≤ 1.5 ULN or endogenous creatinine clearance rate>60ml/min (Cockcroft Gault formula); D. The urine routine test results show that urine protein (UPRO)<2+or 24-hour urine protein quantification<1g;
3. Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%);
4. Coagulation function: International standardized ratio (INR) ≤ 1.5 × ULN and activated partial thromboplastin time ≤ 1.5 × ULN;
5. Pulmonary function: First second forced expiratory volume (FEV1) ≥ 1.2 L, FEV1% ≥ 50%, carbon monoxide diffusion volume (DLCO) ≥ 50%;
6. Other: lipase ≤ 1.5 × ULN (if lipase>1.5) × ULN can be included if there is no clinical or imaging confirmation of pancreatitis; Amylase ≤ 1.5 × ULN (if amylase>1.5 × ULN can be included if there is no clinical or imaging confirmation of pancreatitis; Alkaline phosphatase (ALP) ≤ 2.5ULN.

12.Women of reproductive age should agree that effective contraception must be used during the study period and for 6 months after the study ends; Have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be a non-lactating patient; Men should consent to patients who must use contraception during the study period and for 6 months after the end of the study period;

Exclusion Criteria:

Patients who had any of the following symptoms were excluded from the study:

1. Individuals who are allergic to treatment drugs;
2. Patients who have received standard treatment for liver metastasis colorectal cancer;
3. Previously received anti-tumor therapy or radiation therapy for any malignant tumor;
4. Simultaneously receiving anti-tumor therapies in other clinical trials, including endocrine therapy, bisphosphate therapy, or immunotherapy;
5. Has undergone significant surgical procedures unrelated to colorectal cancer within 4 weeks prior to enrollment, or the patient has not fully recovered from such surgical procedures;
6. Patients with extrahepatic metastasis, unresectable lymph nodes (including portal vein lymph nodes) metastasis, and primary tumor recurrence;
7. Patients whose imaging shows that the tumor has invaded important blood vessels or who have been determined by the researchers to be highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies
8. Within 5 years, subjects have had or co-developed other malignancies requiring active treatment
9. Existence of active autoimmune diseases or immunodeficiency, or a history of autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, pituitary inflammation, vasculitis, nephritis, etc.
10. Individuals who test positive for HIV or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation or allogeneic hematopoietic stem cell transplantation. The following exceptions apply: Patients with a history of autoimmune hypothyroidism who have received thyroid hormone replacement therapy may be included in the study. Patients with type 1 diabetes whose blood sugar can be controlled after treatment with insulin administration scheme can participate in this study.
11. The patient is currently using immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive effects (dosage>10mg/day prednisone or other therapeutic hormones) and continues to use them within 2 weeks prior to enrollment;
12. Patients who have received systemic treatment with high-dose antibiotics within the past 2 weeks;
13. Individuals who have experienced arterial/venous thrombosis events within 6 months prior to the first administration, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral embolism, etc.), deep vein thrombosis, and pulmonary embolism;
14. Cardiovascular diseases with significant clinical significance, including but not limited to acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting surgery within 6 months prior to enrollment; Congestive heart failure: New York Heart Association (NYHA) grade ≥ 2; Ventricular arrhythmia requiring medication treatment (including QTc interval ≥ 450 ms for males and ≥ 470 ms for females); Left ventricular ejection fraction (LVEF)<50%;
15. Active or uncontrolled severe infection (≥ CTCAE5.0 grade 2 infection), including but not limited to hospitalization due to infection complications, bacteremia, or severe pneumonia, unexplained fever>38.5 ℃ before the first administration;
16. Thoracic effusion, pericardial effusion, or ascites with clinical symptoms that require frequent drainage as determined by the researcher;
17. Cirrhosis and active hepatitis; Hepatitis B reference: HBsAg is positive, and HBV DNA exceeds the upper limit of normal value (1000 copies/ml or 500 IU/ml); Patients with past hepatitis B virus (HBV) infection or cured HBV infection (defined as the presence of hepatitis B B core antibody [HBcAb] and the absence of HBsAg, and the normal HBV DNA value detected during the screening period can be included; Hepatitis C reference: HCV antibody positive, and the detection value of HCV virus titer exceeds the upper limit of the normal value/HCV RNA or HCV Ab detection indicates acute and chronic infection;
18. Urine routine indicates urine protein ≥++, and it is confirmed that the 24-hour urine protein quantification is greater than 1.0 g;
19. Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;
20. Patients with pulmonary fibrosis, pneumoconiosis, radiation pneumonia, drug-induced pneumonia, and severe pulmonary dysfunction;
21. Pregnancy (positive pregnancy test before medication) or breastfeeding women;
22. Within 28 days prior to enrollment in this study, surgery (excluding biopsy) was performed or the surgical incision did not fully heal;
23. Received or planned to receive attenuated live vaccines within 4 weeks prior to the first administration;
24. Have received any other investigational drug treatment or participated in other intervention studies within 4 weeks prior to signing the informed consent form;
25. According to the researcher's judgment, patients who are deemed unsuitable for enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-01-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 1 year
  The ration of patients who are evaluated as CR or PR

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 2 years
  Time form treament initation to the first disease progression or death from any cause
Overall survival (OS) | up to 2 years
  Time from treatment initiation until death from any reason
The R0 resection rates The R0 resection rates | 1 year
  The percentage of patients who had a curative (R0) liver metastasectomy following protocol treatment
Adverse events (Safety） | up to 2 years
  adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No